CLINICAL TRIAL: NCT03163615
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Effect of Tibet Rhodiola Capsule on Hypoxia and Cardiovascular Risk Factors in Patients With Obstructive Sleep Apnea: A Pilot Trial
Brief Title: Effect of Tibet Rhodiola Capsule on Hypoxia and Cardiovascular Risk Factors in Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shao-Ping Nie (Other)
Responsible Party: Sponsor-Investigator, Shao-Ping Nie, MD, PhD, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017002
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tibet Rhodiola Capsule (Experimental)
  Interventions: Drug: Tibet Rhodiola Capsule
- Placebo oral capsule (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Tibet Rhodiola Capsule — 4 capsules, po, from admission up to 84 days
  Other Names: Xueyu Hongjingtian Huoli Jiaonang
  Arms: Tibet Rhodiola Capsule
Drug: Placebo oral capsule — 4 capsules, po, from admission up to 84 days
  Arms: Placebo oral capsule

SUMMARY:
The purpose of this study is to evaluate the effect of Tibet Rhodiola Capsule on hypoxia and the cardiovascular risk factors in patients with mild to moderate OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years, males or females;
2. HSAT or PSG testing within recent 3 months;
3. AHI 5-30 and lowest oxygen saturation<85%;
4. Refuse to accept CPAP, Mandibular orthosis device, surgery, or other medications to improve OSA;
5. Written informed consent.

Exclusion Criteria:

1. History of CPAP, Mandibular orthosis device, surgery, or other medications to improve OSA;
2. Significant central sleep apnea;
3. Histories of other sleep disorders: insomnia, chronic sleep deprivation, long-term use of sleeping pills or sedatives, restless legs syndrome;
4. Histories of underlying heart disease (cardiomyopathy, myocarditis, pericarditis or severe valvular disease), cardiogenic shock and heart failure (NYHA or Killip class 3-4), persistent atrial or ventricular arrhythmias;
5. History of myocardial infarction, coronary revascularization, and a known degree of stenosis > 75% of the coronary lesions;
6. Histories of known serious liver dysfunction (ALT or AST levels above 3 times the normal limit), renal insufficiency (GFR<30ml/min), moderate and severe chronic obstructive pulmonary disease, and pulmonary arterial hypertension;
7. Patients with malignant tumors, lymphoma and neuropsychiatric disorders;
8. Patients with major surgery or trauma within 3 months, and active bleeding or cerebrovascular accident within 6 months;
9. History of anemia (hemoglobin<90g/L) or thrombocytopenia (thrombocyte <90×10^9/L);
10. Breastfeeding, pregnant, or potentially fertile women;
11. Patients who have known to be allergic to Tibet Rhodiola Capsule or its components or patients with serious adverse effect;
12. Participation in other clinical trials in recent 3 months;
13. Patients who cannot complete this trial or comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-17 (Actual); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Average oxygen saturation | Change from Baseline to 84±4days
  Average oxygen saturation was assessed by home sleep apnea testing(HSAT)

SECONDARY OUTCOMES:
Lowest saturation | baseline and 84±4days
  Lowest saturation in percentage(%) was assessed by home sleep apnea testing(HSAT)
Percentage of total sleep time associated with saturation lower than 90% (T90SaO2 ) | baseline and 84±4days
  T90SaO2 in percentage(%) was assessed by home sleep apnea testing(HSAT)
AHI | baseline and 84±4days
  AHI was assessed by home sleep apnea testing(HSAT)
Heart rate variability | baseline and 84±4days
  Heart rate variability was assessed by Holter
Coronary flow reserve | baseline and 84±4days
  Coronary flow reserve was assessed by Ultrasonic Cardiogram
Platelet(PLT) count | baseline, 28±2days and 84±4days
  PLT in 10^9/L
Low density lipoprotein-cholesterol(LDL-C) | baseline, 28±2days and 84±4days
  LDL-C in mmol/L
Glycosylated hemoglobin (HbAlc) | baseline and 84±4days
  HbAlc in percentage(%)
Epworth sleepiness scale (ESS) | baseline and 84±4days
  questionnaire
Quality of life scale (WHOQOL-BREF) | baseline and 84±4days
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China